CLINICAL TRIAL: NCT00620464
Title: A Randomized, Double-Blind, Parallel Group, Bioequivalence Study of IMPLANON and Radiopaque IMPLANON
Brief Title: A Bioequivalence Study of IMPLANON and Radiopaque IMPLANON (34528)(P05720)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P05720; 34528
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiopaque Implanon (ro imp) (Active Comparator): The radiopaque rod (Radiopaque Implanon) is similar to the Implanon rod except for the addition of barium sulfate.
  Interventions: Drug: Radiopaque Implanon
- Implanon (imp) (Active Comparator): Implanon® (Org 32222) is a single rod contraceptive implant of 4 cm length and
  2 mm in diameter. Implanon® contains approximately 68 mg etonogestrel (ENG) (Org 3236, 3-ketodesogestrel) dispersed in a matrix of ethylene vinyl acetate (EVA)copolymer, surrounded by an EVA membrane.
  The ENG dose released by Implanon® amounts to about 60-70 μg/day shortly after
  insertion and decreases to about 40 μg/day at the start of the second year, and to about 25-30 μg/day at the end of the third year.
  Interventions: Drug: Implanon (etonogestrel implant)

INTERVENTIONS:
Drug: Radiopaque Implanon — Radiopaque rod for 3 years
  Arms: Radiopaque Implanon (ro imp)
Drug: Implanon (etonogestrel implant) — Implanon (etonogestrel implant) for 3 years
  Arms: Implanon (imp)

SUMMARY:
The primary purpose of this study is to demonstrate the bioequivalence of IMPLANON and Radiopaque IMPLANON.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 but not older than 40 years of age at the time of screening
* Good physical and mental health
* Regular cycles with a usual length between 24 and 35 days
* Body mass index ≥ 18 and ≤ 29
* Willing to give informed consent in writing

Exclusion Criteria:

* Contraindications:

  * known or suspected pregnancy
  * active venous thromboembolic disorder (e.g. deep vein thrombosis,pulmonary embolism)
  * presence or history of severe hepatic disease as long as liver function values have not returned to normal
  * malignancy or pre-malignancy, if sex -steroid-influenced
  * undiagnosed vaginal bleeding
  * hypersensitivity to any of the components of Implanon/Radiopaque Implanon
* Hypertension, i.e. systolic blood pressure >140 mmHg and/or diastolic blood pressure > 90 mmHg.
* A history during pregnancy or during previous use of sex steroids of: jaundice and/or severe pruritus related to cholestasis; gallstone formation; porphyria; systemic lupus erythematosus; haemolytic uraemic syndrome; Sydenham's chorea; herpes gestationis; otosclerosis-related hearing loss
* Present use or use during 2 months prior to the start of Implanon/Radiopaque Implanon of one of the following drugs: phenytoin, phenobarbital, primidone, carbamazepine, rifampicin, oxcarbazepine, topiramate, felbamate, ritonavir, nelfinavir, griseofulvin or the herbal remedy St John's wort.
* Administration of investigational drugs within 2 months prior to the start of Implanon/Radiopaque Implanon

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2005-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

REFERENCES:
- [Derived] Schnabel P, Merki-Feld GS, Malvy A, Duijkers I, Mommers E, van den Heuvel MW. Bioequivalence and x-ray visibility of a radiopaque etonogestrel implant versus a non-radiopaque implant: a 3-year, randomized, double-blind study. Clin Drug Investig. 2012 Jun 1;32(6):413-22. doi: 10.2165/11631930-000000000-00000. PMID 22540269

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiopaque Implanon (ro Imp) | Implanon (Imp)
Started | 52 | 56
Completed | 32 | 32
Not Completed | 20 | 24
Not completed — Adverse Event | 15 | 17
Not completed — Lost to Follow-up | 1 | 1
Not completed — Planning Pregnancy | 1 | 4
Not completed — Personal | 2 | 2
Not completed — Used prohibited medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiopaque Implanon (ro Imp) | Implanon (Imp) | Total
Number analyzed (Participants) | 52 | 56 | 108
Age, Customized [Number; unit: participants] — Despite the protocol inclusion criteria, one patient was enrolled who was older than 40 years old. The subject was 43 years old.
  participants
    18-20 years | 11 | 12 | 23
    21-25 years | 9 | 18 | 27
    26-30 years | 15 | 10 | 25
    31-35 years | 6 | 12 | 18
    36-40 years | 10 | 4 | 14
    41-45 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 56 | 108
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence of Implanon® and Radiopaque Implanon.
Description: Bioequivalence testing was performed based on serum etonogestrel AUC0-6months, AUC0-24months, and AUC0-36months. Bioequivalence was to be concluded when the 90% confidence limits of AUC0-6months, AUC0-24months, and AUC0-36months were fully contained within the acceptance range of 0.80-1.25.
  AUC0-6months (Area under the curve from zero to six months).
  AUC0-24months (Area under the curve from zero to 24 months).
  AUC0-36months (Area under the curve from zero to 36 months).
Time Frame: 3 years
Population: 103 subjects were pharmacokinetically evaluable. Subjects were excluded from PK evaluation for use of protocol-prohibited steroidal medication during the trial or contraceptives within 1 week prior to Implanon insertion, or because their pre-insertion ENG concentration was not proven to be below the Lower Limit of Quantification (LLOQ)
Measure: Mean (Full Range); unit: pg•month/mL
Arm/Group | Radiopaque Implanon (ro Imp) | Implanon (Imp)
Number analyzed (Participants) | 50 | 53
pg•month/mL
  AUC (0-6 months) (n=46 ro imp; n=46 imp) | 2296 [1320 to 4033] | 2290 [1386 to 3773]
  AUC (0-24 months) (n=37 ro imp; n=32 imp) | 5954 [3687 to 10080] | 6131 [3625 to 11500]
  AUC (0-36 months) (n=32 ro imp; n=30 imp) | 7667 [4702 to 12620] | 7819 [4843 to 15114]
Statistical Analysis 1: Comparison: Radiopaque Implanon (ro Imp) vs Implanon (Imp); Test type: Superiority or Other; p = 0.05, Bioequivalence Testing — Applies to all parameters

2. Primary Outcome: Bioequivalence of Implanon® and Radiopaque Implanon
Description: Bioequivalence testing was performed based on serum etonogestrel Cmax. Bioequivalence was to be concluded when the 90% confidence limits of Cmax were fully contained within the acceptance range of 0.80-1.25.
  Cmax (pg/mL): Peak concentration.
Time Frame: 3 years
Population: All-Subjects-Pharmacokinetically-Evaluable consisted of 103 subjects.Subjects excluded from PK evaluation due to age, use of by protocol prohibited steroidal medication during trial and contraceptives within one week prior to Implanon insertion and their pre-insertion ENG concentration was not proven to be below Lower Limit Of Quantification (LLOQ)
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Radiopaque Implanon (ro Imp) | Implanon (Imp)
Number analyzed (Participants) | 50 | 53
pg/mL | 1200 [509 to 3030] | 1145 [317 to 3100]
Statistical Analysis 1: Comparison: Radiopaque Implanon (ro Imp) vs Implanon (Imp); Test type: Superiority or Other; p <= 0.05, Bioequivalence Testing

ADVERSE EVENTS:
Groups:
- Implanon: Implanon® (Org 32222) is a single rod contraceptive implant of 4 cm length and 2 mm in diameter. Implanon® contains approximately 68 mg etonogestrel (ENG) (Org 3236, 3-ketodesogestrel) dispersed in a matrix of ethylene vinyl acetate (EVA)copolymer, surrounded by an EVA membrane.
  The ENG dose released by Implanon® amounts to about 60-70 μg/day shortly after insertion and decreases to about 40 μg/day at the start of the second year, and to about 25-30 μg/day at the end of the third year.
- Radiopaque Implanon: The radiopaque rod (Radiopaque Implanon) is similar to the Implanon rod except for the addition of barium sulfate.
Arm/Group | Implanon | Radiopaque Implanon
Serious Adverse Events (participants affected / at risk) | 6/56 | 4/52
Other Adverse Events (participants affected / at risk) | 54/56 | 48/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanon (N=56) | Radiopaque Implanon (N=52)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vertebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mammoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Scar excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanon (N=56) | Radiopaque Implanon (N=52)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (7)
Nausea (Gastrointestinal disorders) | 8 (9) | 6 (8)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 3 (5) | 2 (2)
Hangover (General disorders) | 2 (3) | 3 (3)
Implant site haematoma (General disorders) | 16 (16) | 16 (16)
Implant site pain (General disorders) | 6 (9) | 4 (5)
Seasonal allergy (Immune system disorders) | 3 (5) | 2 (2)
Cystitis (Infections and infestations) | 4 (4) | 8 (9)
Gastroenteritis (Infections and infestations) | 4 (4) | 6 (10)
Influenza (Infections and infestations) | 14 (23) | 12 (27)
Nasopharyngitis (Infections and infestations) | 14 (21) | 18 (42)
Sinusitis (Infections and infestations) | 3 (4) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 2 (3) | 4 (6)
Vulvovaginal mycotic infection (Infections and infestations) | 7 (8) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 5 (6)
Weight decreased (Investigations) | 4 (4) | 1 (1)
Weight increased (Investigations) | 8 (8) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 11 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 5 (6) | 5 (5)
Headache (Nervous system disorders) | 15 (38) | 14 (39)
Amenorrhoea (Reproductive system and breast disorders) | 6 (7) | 3 (3)
Breast pain (Reproductive system and breast disorders) | 4 (5) | 4 (5)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 4 (6)
Dysmenorrhoea (Reproductive system and breast disorders) | 4 (9) | 6 (19)
Genital haemorrhage (Reproductive system and breast disorders) | 23 (52) | 24 (69)
Metrorrhagia (Reproductive system and breast disorders) | 9 (11) | 9 (10)
Oligomenorrhoea (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 5 (8) | 3 (4)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 3 (4)
Vaginal discharge (Reproductive system and breast disorders) | 3 (5) | 3 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 18 (63) | 21 (151)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (8)
Acne (Skin and subcutaneous tissue disorders) | 18 (32) | 11 (22)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All investigator publications must be based on data validated and released by sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to sponsor, at least six weeks ahead of estimated publication or presentation, for consent. In the event that no response is received within six weeks after submission, the investigator may use the submitted data.